CLINICAL TRIAL: NCT01184495
Title: Comparison of the Efficacy of Erythropoietin Produced in the Institute of Technology in Immunobiology of the Oswald Cruz Foundation (BioMaguinhos/FioCruz/MS) and Erythropoietin Industrialized in Patients With Chronic Renal Failure
Brief Title: Efficacy Study of Two Formulations of Erythropoietin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Rio Grande do Sul State Health Department - SES/RS (Other Government); Oswaldo Cruz Foundation (Other)
Responsible Party: Principal Investigator, Paulo Dornelles Picon, MhD, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-168
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Comparison of the Efficacy of Two Formulations of Epoetin in Patients Undergoing Hemodialysis
Keywords: Erythropoietin; Chronic renal failure; Hemodialysis; Anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epoetin Bio-Manguinhos (Experimental)
  Interventions: Drug: Epoetin Alfa-BioManguinhos
- EPO-BioSimilar (Active Comparator): Subcutaneous administration of EPO-BioSimilar
  Interventions: Drug: Epoetin Alfa-BioSimilar

INTERVENTIONS:
Drug: Epoetin Alfa-BioManguinhos — Subcutaneous administration of EPO-BioManguinhos
  Arms: Epoetin Bio-Manguinhos
Drug: Epoetin Alfa-BioSimilar — Subcutaneous administration of EPO-BioSimilar
  Arms: EPO-BioSimilar

SUMMARY:
A double-blind, randomized trial aimed to compare the efficacy of two formulations of erythropoietin in patients with chronic renal failure on hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* We included adult patients with chronic renal failure on hemodialysis for more than three months at the Dialysis Unit of the Department of Nephrology, HCPA and the Center for Dialysis and Transplant (CDT), characterized as as patients on chronic regular dialysis procedure. Patients already in use of EPO for at least three months, only those taking the drug by subcutaneous and agreed to participate in the study.

Patients using different doses of EPO were included, but these were distributed across the treatment groups by randomization stratum dose of EPO, to ensure even distribution of patients in both groups.

It was considered that patients with HIV or AIDS who were in treatment for the disease with proper clinical management would be eligible for the study (as exemplified by patients with HIV or AIDS approved for inclusion on the waiting list for cadaveric kidney transplantation) .

Patients with a history of cancer or already treated in the oncological standpoint, and no signs of disease activity could be included.

Exclusion Criteria:

* Patients who had other causes of anemia defined for maintenance, for example, patients with liver cirrhosis, with a history of gastrointestinal bleeding, patients with chronic Gastro Intestinal, Genital or Urinary bleeding or other sites were excluded. Similarly patients with AIDS without treatment, hemolytic anemia, pancytopenia, thalassemia, sickle cell anemia, myelodysplasia, multiple myeloma or other cancers or inflammatory arthritis. There was also no inclusion of patients with intolerance or allergy to iron parenterally, patients without adherence to dialysis or with chronic inadequate dialysis blood flow of vascular access persistently below 250 mL / min, kt / v, as a measure of efficiency of hemodialysis, persistently <1.2) or frequent hospitalizations considered as possible causes of inadequate response to erythropoietin.

We excluded patients with mental illness or condition that prevents the free consent and signature of informed consent, as well as previous reports of serious adverse effects to the drugs studied.

Criteria for withdrawal from the clinical trial: a view of the high morbidity of hemodialysis patients, expressed by frequent hospital clinics, it was found that patients in the study would not be withdrawn from the study due to hospitalization, provided that: the hospital did not involve surgery (except vascular access surgery or hospitalization in the intensive care unit or equivalent, or that represent otherwise, a loss of patient follow-up or co-interventions in the treatment of anemia of these).

Were withdrawn from the study patients who required blood transfusion because they have severe anemia or intervention unrelated to the usual treatment of anemia in hemodialysis patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2008-04; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin Level in blood | Monthly assessment of the levels of hemoglobin in blood at baseline and monthly for six months
  The evaluation of the efficacy between different formulations of recombinant EPO: the one produced by Bio-Manguinhos and produced by private industry was observed in response to EPO as measured by levels of hemoglobin (Hb) results. The mean Hb of the two groups were compared, as well as the variation observed in both groups over time follow-up (six months).

SECONDARY OUTCOMES:
Safety | Monthly assessment of adverse events
  Assessing the safety of the formulation produced by Bio-Manguinhos was performed by comparing the rate of adverse events related to the use of recombinant EPO in the two study groups

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Dornelles Picon, Principal Investigator — Hospital de Clinicas de Porto Alegre

REFERENCES:
- [Derived] Picon PD, Pribbernow SC, Prompt CA, Schacher SC, Antunes VV, Mentz BP, Oliveira FL, Souza CM, Schacher FC. Randomized double-blind clinical trial of a new human epoetin versus a commercially available formula for anemia control in patients on hemodialysis. Clinics (Sao Paulo). 2014 Aug;69(8):547-53. doi: 10.6061/clinics/2014(08)08. PMID 25141114